CLINICAL TRIAL: NCT04024072
Title: Multi-Center, Randomized, Double-Masked, Active Controlled, Parallel Group Study to Compare Perrigo's Brinzolamide Ophthalmic Suspension 1% to Azopt® in the Treatment of Primary Open Angle Glaucoma or Ocular Hypertension in Both Eyes
Brief Title: To Compare the Safety and Efficacy of Perrigo's Product to an FDA Approved Product for the Treatment of Glaucoma or Ocular Hypertension in Both Eyes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-19-001
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perrigo active (Experimental): Test product
  Interventions: Drug: Brinzolamide 1% ophthalmic suspension
- Reference active (Active Comparator): Azopt ophthalmic suspension
  Interventions: Drug: Azopt 1% Ophthalmic Suspension

INTERVENTIONS:
Drug: Brinzolamide 1% ophthalmic suspension — Test product
  Arms: Perrigo active
Drug: Azopt 1% Ophthalmic Suspension — Reference product
  Arms: Reference active

SUMMARY:
To compare the safety and efficacy of Perrigo's product to an FDA approved product in the treatment of Primary Open Angle Glaucoma or Ocular Hypertension in Both Eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant females aged at least 18 years with chronic open angle glaucoma or ocular hypertension in both eyes
2. Subject requires treatment of both eyes and is able to discontinue use of all ocular hypotensive medication(s) or switch ocular hypotensive medications and undergo appropriate washout period.
3. Adequate wash-out period prior to baseline of any ocular hypotensive medication.
4. Baseline (Day 0/hour 0) pressure ≥ 22 mm Hg and ≤ 34 mm Hg in each eye and any asymmetry of pressure between the eyes no greater than 5 mm Hg.
5. Baseline best corrected visual acuity equivalent to 20/200 or better in each eye

Exclusion Criteria:

1. Females who are pregnant, breast feeding, or planning a pregnancy.
2. Females of childbearing potential who do not agree to utilize an adequate form of contraception
3. Current, or past history of, severe hepatic or renal impairment
4. Current, or history within two months prior to baseline of, significant ocular disease, e.g., corneal edema, uveitis, ocular infection, or ocular trauma in either eye
5. Current corneal abnormalities that would prevent accurate readings with the Goldmann applanation tonometer
6. Functionally significant visual field loss
7. Contraindication to brinzolamide or sulfonamide therapy or known hypersensitivity to any component of brinzolamide or sulfonamide therapy
8. Use at any time prior to baseline of an intraocular corticosteroid implant
9. Use within one week prior to baseline of contact lens
10. Use within two weeks prior to baseline of: 1) topical ophthalmic corticosteroid, or 2) topical corticosteroid
11. Use within one month prior to baseline of: 1) systemic corticosteroid or 2) high-dose salicylate therapy
12. Use within six months prior to baseline of intravitreal or subtenon injection of ophthalmic corticosteroid
13. Having undergone within six months prior to baseline any other intraocular surgery (e.g., cataract surgery)
14. Having undergone within twelve months prior to baseline refractive surgery, filtering surgery, or laser surgery for pressure reduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- James D. Branch Ophthalmology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perrigo Active | Reference Active
Started | 249 | 246
Completed | 247 | 237
Not Completed | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perrigo Active | Reference Active | Total
Number analyzed (Participants) | 249 | 246 | 495
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 96 | 194
  >=65 years | 151 | 150 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.85) | 65.6 (11.12) | 65.7 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 132 | 277
  Male | 104 | 114 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 31 | 56
  Not Hispanic or Latino | 223 | 215 | 438
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 81 | 84 | 165
  White | 161 | 155 | 316
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Iris Color [Count of Participants; unit: Participants]
  Right eye: Dark | 158 | 163 | 321
  Right eye: Light | 91 | 83 | 174
  Left eye: Dark | 158 | 162 | 320
  Left eye: Light | 91 | 84 | 175

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intra-ocular Pressure
Description: mean change in intra-ocular pressure of both eyes at four time points : at approximately 8:00 a.m. (hour 0; before the morning drop) and approximately 10:00 a.m. (hour 2) on Day 14 (Week 2) and Day 42 (Week 6) visits.
Time Frame: 6 weeks
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Perrigo Active | Reference Active
Number analyzed (Participants) | 228 | 219
mmHG
  8AM Day 14 | -4.25 (2.713) | -3.80 (2.719)
  10AM Day 14 | -4.22 (2.722) | -4.00 (2.756)
  8AM Day 42 | -4.43 (2.967) | -4.20 (2.591)
  10AM Day 42 | -4.05 (2.961) | -4.06 (2.842)
Statistical Analysis 1: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — 8AM Day 14; Mean Difference (Net) = -0.46, 95% CI 2-sided [-0.93 to 0.01]
Statistical Analysis 2: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — 10AM Day 14; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.70 to 0.24]
Statistical Analysis 3: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — 8AM Day 42; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.74 to 0.27]
Statistical Analysis 4: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — 10AM Day 42; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.51 to 0.51]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 46
Arm/Group | Perrigo Active | Reference Active
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/246
Serious Adverse Events (participants affected / at risk) | 0/249 | 1/246
Other Adverse Events (participants affected / at risk) | 32/249 | 36/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perrigo Active (N=249) | Reference Active (N=246)
Upper respiratory tract infection (Infections and infestations) | NA | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perrigo Active (N=249) | Reference Active (N=246)
vision blurred (Eye disorders) | 9 (9) | 15 (15)
Dysgeusia (Nervous system disorders) | 23 (23) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04024072/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04024072/SAP_001.pdf